CLINICAL TRIAL: NCT00552981
Title: Effectiveness of Local Application of Warm Air in Patients With Common Cold (HELI Study)
Acronym: HELI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Karl and Veronica Carstens Foundation (Other)
Responsible Party: Principal Investigator, Claudia M. Witt, Prof. Dr. med., Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HELI-2007
Record Dates: First submitted 2007-11-01; First posted 2007-11-02 (Estimated); Last update posted 2012-07-10 (Estimated); Status verified 2012-07

CONDITIONS: Common Cold
Keywords: common cold; Finnish sauna; rct
MeSH Terms: conditions — Common Cold

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator)
  Interventions: Procedure: inhalation of warm air in a Finnish sauna
- 2 (Sham Comparator)
  Interventions: Procedure: inhalation of ambient air in a Finnish sauna

INTERVENTIONS:
Procedure: inhalation of warm air in a Finnish sauna — three times on three following days, each 2-3 minutes
  Arms: 1
Procedure: inhalation of ambient air in a Finnish sauna — three times on three following days, each 2-3 minutes
  Arms: 2

SUMMARY:
In a randomized controlled trial, the investigators include patients with beginning symptoms of a common cold and compare two interventions:

1. the inhalation of warm air for inducing a warming of the throat and
2. the inhalation of ambient air as control. As outcome the effect on symptoms and duration of the common cold will be assessed. The interventions will consist of visits with a duration of 2-3 minutes on three following days in a Finnish sauna. Patients will be fully dressed.

ELIGIBILITY:
Inclusion Criteria:

* symptom duration between 2 and 24 hours
* at least two of the ten following symptoms: cough, headache, hoarseness, muscle ache, nasal drainage, nasal congestion, scratchy throat, sore throat, sneezing, and fever
* no usage of medication bought in a pharmacy
* informed consent

Exclusion Criteria:

* fever >38.5°C
* systolic blood pressure below 100 mmHg or above 160 mmHg
* severe chronic disease, which makes study participation impossible
* pregnancy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 157 (Actual)
Dates: Start 2007-11; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Symptom Score for Common Cold | Area under the curve day 2 to 7

SECONDARY OUTCOMES:
Usage of medication against common cold | Day 1 to 7
generalized feeling ill on a numeric rating scale 0-10, | Day 1, 2, 3, 5 and 7
safety (adverse events and serious adverse events) | 1 to 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Claudia M. Witt, MD, Principal Investigator — Institute for Social Medicine, Epidemiology, and Health Economics, Charité University Medical Center, Berlin, Germany
Locations (1):
- Institute for Social Medicine, Epidemiology, and Health Economics, Charité University Medical Center, Berlin, Germany

REFERENCES:
- [Result] Pach D, Knochel B, Ludtke R, Wruck K, Willich SN, Witt CM. Visiting a sauna: does inhaling hot dry air reduce common cold symptoms? A randomised controlled trial. Med J Aust. 2010 Dec 6-20;193(11-12):730-4. doi: 10.5694/j.1326-5377.2010.tb04127.x. PMID 21143077